CLINICAL TRIAL: NCT02022865
Title: Correlation Between Inflammatory Markers in Gingival Crevicular Fluid, Serum and Amniotic Fluids in Periodontal Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Polak David, senior physician, Hadassah Medical Organization
Other Study IDs: HMO-12-0412
Record Dates: First submitted 2013-12-11; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Periodontal Disease; Adverse Pregnancy Outcome
Keywords: periodontitis; cytokines; adverse pregnancy outcome
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — gingival crevicular fluid, serum, aminiotic fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- periodontitis patients: according to american academy of periodontology classification of periodontal diagnosis.
- healthy periodontium: according to american academy of periodontology classification of periodontal diagnosis.

SUMMARY:
The main causes of adverse pregnancy outcome(s) are reported to be maternal infection and placental, foetal, or uterine pathosis. Maternal infection and placental pathosis appear to be the most important causal factors, possibly causing pre-term labour, premature pre-term membrane rupture, or result in medically induced pregnancy interruption. There are reports of a link between poor maternal periodontal health and composite adverse pregnancy outcome of pre-term low birth weight (PLBW). however, the reason for such correlation is still not clear.

In the current study the investigators will try to follow a possible path between periodontal infection and uterus physiology, by signaling out inflammatory markers that may leak from the gingival fluid into the serum and from there to the amniotic fluid.

the investigators will collect GCF, serum and amniotic fluid from patients undergoing elective amniocentesis and analyse inflammatory markers in the collected samples.

DETAILED DESCRIPTION:
Globally, over 4 million babies die within the first 4 weeks of life and a third of these are secondary to pre-term birth. In the United States, pre-term birth is the second leading cause of neonatal mortality. The US pre-term birth (<37 weeks) rate rose to 12.8% in 2006, an increase of 21% since 1990 and the rate of low birthweight (<2500 g) rose to 8.3% in 2006, an increase of 19% since 1990. Neurological disorders, such as cerebral palsy, which is often combined with mental disability, epilepsy, and cognitive impairment, are of special concern for survivors of pre-term birth. Even though pre-term birth occurs in only a small proportion of the infant population, its societal and personal health impact is considerable because of its disproportionately high perinatal morbidity, mortality, and need for costly medical care. However, it is very disappointing that to date, interventions to prevent pre-term birth have proven to be almost universally ineffective.

The main causes of adverse pregnancy outcome(s) are reported to be maternal infection and placental, fetal, or uterine pathosis. Maternal infection and placental pathosis appear to be the most important causal factors, but each can cause pre-term labour, premature pre-term membrane rupture, or result in medically induced pregnancy interruption. Prominent risk factors for pre-term birth include history of previous pre-term birth, demographic characteristics, periodontal disease, and behavioral factors such as tobacco use.

Offenbacher et al. were the first to report a link in humans between poor maternal periodontal health and composite adverse pregnancy outcome of pre-term low birth weight (PLBW). They reported that women with periodontal disease were much more likely than periodontally healthy women to experience pre-term and low birth weight infants (OR=7.5 for all PLBW cases; OR=7.9 for primiparous PLBW cases). Pro-inflammatory mediators generated within the diseased periodontal tissue may affect the maternal-foetal unit. When present in the amniotic fluid, chronic high levels of cytokines and prostaglandins may lead to intra-uterine growth restriction (IUGR), spontaneous pre-term labour, premature rupture of membranes, and pre-term birth. Several studies report associations of adverse pregnancy outcome with higher gingival crevicular fluid levels of PGE2 and IL-1β and elevated amniotic fluid concentrations of PGE2, IL-1β and IL-8 Dörtbudak. It is possible that IL-6 produced in inflamed periodontal tissues can affect the foetal membranes and cause pre-term uterine contractions. There is evidence that the gingival crevicular fluid levels of IL-6 are higher in gingivitis and periodontitis compared with healthy controls.

Bacteria activate cell-mediated immunological responses, leading to the production and release of cytokines, including interleukin-1 (IL-1), IL-6, tumor necrosis factor-α (TNF-α), prostaglandins, or endotoxins such as lipopolysaccharides, which may precipitate pre-term labour if they reach the foeto-placental unit. Endotoxin or lipopolysaccharide of Gram-negative bacteria may be detected in biological fluids of sterile compartments such as the amniotic cavity. Administration of endotoxin to pregnant animals results in embryo resorption, pre-term labour, and foetal death. A higher risk of spontaneous pre-term delivery has been associated with genetically driven excessive amniotic fluid IL-Iβ or with a disturbance of bioavailability and/or bio-response of this cytokine, which is central to the pro-inflammatory reaction to infectious stimulants. The foetus also has a role in pre-term birth; the foetus recognizes a hostile intrauterine environment and may precipitate labour by premature activation of the foetal-placental parturition pathway.

The causality relationship between periodontal disease and inflammatory mediators' presence in the amnionic fluid was not tested to date. In the present study the investigators aim to investigate the correlation between inflammatory mediators in the serum and their presence in the amniotic fluid. The investigators will further investigate the correlation of the above results with pregnancy outcome (gestation age, foetal weight and health, etc.).

Israel amniocentesis in healthy women is very common. The cellular fraction in the sampled amniotic fluid is used for the amniocentesis test, while the supernatant is discarded. For the present study the investigators aim to use the supernatants of amniocentesis tests done on healthy women (age 21-45) as well as serum. Using ELISA we will quantify the levels of inflammatory markers such as IL-6, TNFα and IL-1β. The investigators will also test the presence of endotoxin and perio-pathogens DNA in the serum and amnionic fluid. Follow-up on data regarding gestational outcome will be also collected.

participants will be followed for the duration of hospital stay, an expected average of 5 weeks

ELIGIBILITY:
Inclusion Criteria:

* age 18-45
* single fetus pregnancy
* at least 20 teeth present

Exclusion Criteria:

* high risk pregnancy
* alcohol consumption
* smoking
* pregnancy diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy pregnant women, undergoing elective amniocentesis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
cytokines levels | analysed at the end of sample collection. participants will be followed for the duration of pregnancy, an expected average of 5 months
  Using ELISA we will quantify the levels of inflammatory markers such as IL-6, TNFα and IL-1β.

SECONDARY OUTCOMES:
presence of endotoxin and perio-pathogens DNA in the serum and amnionic fluid | analysed at the end of sample collection. participants will be followed for the duration of pregnancy, an expected average of 5 months
  We will also test the levels of endotoxin and perio-pathogens DNA in the serum and amniotic fluid using real time PCR and ELISA. Measures are a composite outcome measure consisting of multiple measures (results to be reported as a single value for each Arm/Group).

REFERENCES:
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Offenbacher S, Jared HL, O'Reilly PG, Wells SR, Salvi GE, Lawrence HP, Socransky SS, Beck JD. Potential pathogenic mechanisms of periodontitis associated pregnancy complications. Ann Periodontol. 1998 Jul;3(1):233-50. doi: 10.1902/annals.1998.3.1.233. PMID 9722707